CLINICAL TRIAL: NCT06637007
Title: Single Arm, Open Phase II Clinical Trial of Chidamide Combined With AK112 for Second-line and Advanced Bone and Soft Tissue Sarcoma
Brief Title: Phase II Clinical Trial of Chidamide Combined With AK112 for Second-line and Advanced Bone and Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanxi Province Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: zlyygcp; zlyygcp (Other: Shanxi Cancer Hospital)
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Sarcoma,Soft Tissue; Sarcoma; Sarcoma of Bone
MeSH Terms: conditions — Sarcoma; Osteosarcoma | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chidamide Tablets combined with AK112 (Experimental): 1. Medication dosage：Chidamide Tablets（30mg,Twice a week，po），AK112（Once every 3 weeks）.
     If you experience any discomfort during the medication process, please inform your responsible doctor in a timely manner. He/she will provide appropriate treatment based on the severity of the reaction. In severe cases, the dosage of medication will be adjusted until it is stopped.
  2. Medication method: The interval between two oral doses of Xidabenzamide should not be less than 3 days (such as Monday and Thursday, Tuesday and Friday, Wednesday and Saturday, etc.), and should be taken 30 minutes after breakfast. During the research process and before the end of medication, the responsible doctor will conduct physical and laboratory examinations on you in accordance with the experimental protocol to evaluate the impact of the experimental drug on you.
  Interventions: Drug: Chidamide Tablets combined with AK112

INTERVENTIONS:
Drug: Chidamide Tablets combined with AK112 — Chidamide Tablets 30mg/day, po.Bid; AK112（10mg/kg or 20mg/kg）, ivgtt, Q3W.
  Other Names: AK112

SUMMARY:
Evaluation of the efficacy and safety of Xidabenzamide combined with AK112 for advanced bone and soft tissue sarcoma of second-line and above.

DETAILED DESCRIPTION:
Evaluation of the efficacy and safety of Xidabenzamide combined with AK112 for advanced bone and soft tissue sarcoma of second-line and above.

Main objective: To explore the objective response rate (ORR) and progression free survival (PFS) of Xidabenzamide combined with AK112 for disease stability in advanced bone and soft tissue sarcoma of second-line and above Secondary objective: To explore the overall survival (OS), quality of life (QOL), safety, and tolerability indicators of Xidabenzamide combined with AK112 for advanced bone and soft tissue sarcoma of second-line and above.

ELIGIBILITY:
Inclusion Criteria:

* The patient voluntarily participated in this study and signed an informed consent form；
* All advanced bone and soft tissue sarcomas diagnosed by pathology have at least one measurable lesion according to RECIST 1.1 criteria, mainly including synovial sarcoma, smooth muscle sarcoma, vascular sarcoma, undifferentiated pleomorphic sarcoma/malignant fibrous histiocytoma, liposarcoma, fibrosarcoma, clear cell sarcoma, epithelioid sarcoma, malignant peripheral nerve sheath tumor, undifferentiated sarcoma, rhabdomyosarcoma, protuberant skin fibrosarcoma, Ewing's sarcoma/primary neuroectodermal tumor, connective tissue proliferative small round cell tumor, inflammatory myofibroblastic sarcoma, malignant solitary fibroadenoma, chondrosarcoma, osteosarcoma. Except for the following types: malignant mesothelioma, acinar soft tissue sarcoma, gastrointestinal stromal tumor, and extra bone mucinous chondrosarcoma;
* Patients with advanced bone and soft tissue sarcoma who experience disease progression or failure after first-line standard treatment;
* 18~75 years old; ECOG PS score: 0-1 points; Expected survival period exceeding 3 months;
* Adequate organ and bone marrow function, no severe hematopoietic dysfunction, heart, lung, liver, kidney, thyroid dysfunction, or immunodeficiency (no blood transfusion, granulocyte colony-stimulating factor, or other related medical support received within 14 days prior to the use of the study drug)；
* The main organ function meets the following criteria within 7 days before treatment:

  1. Blood routine examination standard (without blood transfusion within 14 days)：

     * hemoglobin（HB）≥90g/L；

       * Absolute Neutrophil Count（ANC）≥1.5×109/L；

         * platelet（PLT）≥80×109/L。
  2. Biochemical tests must meet the following standards：

     * total bilirubin（TBIL）≤1.5 upper limit of normal (ULN) ；

       * Alanineaminotransferase（ALT）and Aspartic transaminaseAST≤2.5 ULN，If accompanied by liver metastasis, ALT and AST≤5 ULN；

         * Serum creatinine（SCr）≤1.5 ULN or Creatinine clearance rate(CCr)≥60ml/min；
  3. Doppler ultrasound evaluation：Left ventricular ejection fraction (LVEF) ≥ Low limit of normal (50%)。
* Thyroid Stimulating Hormone（TSH）or Free Thyroxine（FT4）or Free triiodothyronine（FT3）all within the normal range of ± 10%.
* Women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, birth control pills, or condoms) during the study period and within 6 months after the end of the study; Serum or urine pregnancy test negative within 7 days prior to enrollment in the study, and must be non lactating.
* patient; Men should agree to patients who must use contraception during the study period and within 6 months after the end of the study period.

Exclusion criteria: Patients with any of the following conditions will not be included in this study

* Patients who have previously used sildenafil or other histone deacetylase inhibitors;
* Previously received treatment with immune checkpoint inhibitors (PD-1, PD-L1, CTLA-4, etc.);
* Other malignant tumors that have occurred or are currently present within the past 5 years, except for cured cervical carcinoma in situ, non melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor infiltrating basement membrane)];
* Received systemic anti-tumor therapy, including chemotherapy, immunotherapy, and biological therapy (such as tumor vaccines, cytokines, or growth factors that control cancer), within 28 days before starting the research treatment;
* Have received Chinese herbal medicine or traditional Chinese patent medicines and simple preparations with anti-tumor indications within 7 days before starting the research treatment;
* Planned systemic anti-tumor therapy within 4 weeks prior to enrollment or during the study medication period, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or use of mitomycin C within 6 weeks prior to receiving experimental drug treatment). Expanded field radiation therapy (EF-RT) was performed within 4 weeks prior to enrollment, or limited field radiation therapy was performed within 2 weeks prior to grouping to assess tumor lesions;
* Accompanied by pleural effusion or ascites, causing respiratory syndrome (≥ CTC AE grade 2 respiratory distress [grade 2 respiratory distress refers to shortness of breath during light activity; affects instrumental daily activities]);
* Unrelieved toxic reactions above CTC AE (4.01) grade 1 caused by any previous treatment, excluding hair loss;
* Patients with brain metastases accompanied by symptoms or symptom control time less than 2 months;
* Patients with any severe and/or uncontrolled illnesses, including:

  1. Patients with poor blood pressure control (systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 100 mmHg);
  2. Suffering from grade I or above myocardial ischemia or myocardial infarction, arrhythmia (including QTC ≥ 480ms), and grade ≥ 2 congestive heart failure (NYHA classification);
  3. Active or uncontrolled severe infections (≥ CTC AE level 2 infection);
  4. Cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral therapy;
  5. Renal failure requires hemodialysis or peritoneal dialysis;
  6. Individuals with a history of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
  7. Poor control of diabetes (FBG>10mmol/L);
  8. Urine routine shows urinary protein ≥++and confirms 24-hour urinary protein quantification>1.0 g;
  9. Patients with epileptic seizures who require treatment;
* Received major surgical treatment, open biopsy, or significant traumatic injury within 28 days prior to enrollment;
* Patients with any signs or medical history of bleeding, regardless of the severity; Patients who have experienced any bleeding or bleeding events ≥ CTCAE grade 3 within the first 4 weeks of enrollment, with unhealed wounds, ulcers, or fractures;
* Individuals who have experienced arterial/venous thrombotic events within the past 6 months, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis, and pulmonary embolism;
* Patients with active ulcers, intestinal perforation, and intestinal obstruction;
* Individuals with a history of abuse of psychotropic drugs who are unable to quit or have mental disorders;
* Participated in clinical trials of other anti-tumor drugs within 28 days prior to enrollment;
* According to the researchers' judgment, there are accompanying diseases that seriously endanger patient safety or affect the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy of the investigational drug will be determined by the objective tumor evaluation conducted by the research center based on the RECIL 2017 lymphoma efficacy evaluation criteria | Baseline and testing every 6 weeks
  The imaging evaluation methods for tumors are PET/CT, MR, or CT, but the evaluation methods, machines, and technical parameters should be consistent throughout the entire study period. The imaging results are interpreted by researchers or radiologists from each research center. If tumor evaluation has been conducted within 21 days before enrollment and the same methods and machines are used in the same hospital, it can be used as a baseline tumor evaluation. Baseline tumor evaluation should include the nasal cavity, chest, abdomen, pelvic cavity, and any other suspected tumor lesions. If there are clinical indications, appropriate methods can be used to examine any other known or suspected disease site, such as cranial MRI or bone scan.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, Study Director — Shanxi Province Cancer Hospital
Locations (1):
- Shanxi Cancer Hospital, Taiyuan, Shanxi, China